CLINICAL TRIAL: NCT06705712
Title: A Preconception Cohort Study of Physical Activity, Fertility, and Spontaneous Abortion - Including a Randomized Controlled Trial.
Brief Title: Physical Activity, Fertility, and Spontaneous Abortion in Danish Couples Trying to Conceive
Acronym: SF/Activity
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1-10-72-174-23
Record Dates: First submitted 2024-10-29; First posted 2024-11-26 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2024-06

CONDITIONS: Fertility; Fecundability; Time-to-Pregnancy; Spontaneous Abortion; Pregnancy Outcome; Pregnancy Complications
Keywords: Exercise; Physical activity; Sedentary behaviour; Fertility; Spontaneous abortion; Preconception care; Fecundability; Time to pregnancy
MeSH Terms: conditions — Abortion, Spontaneous; Pregnancy Complications; Motor Activity

STUDY DESIGN:
Intervention Model Description: SnartForældre/Activity is designed as a two-armed randomized controlled trial, including 530 women, who are trying to conceive. Included participants will be randomized in a 1:1 ratio to an intervention group or a control group. The participates are followed during preconception for up to a year or until they conceive. The participants who conceive during the study period are followed during their first trimester of the pregnancy or until they experience a pregnancy loss. Collection of data for assessment of the outcomes was through bimonthly follow-up questionnaires linked with registry data. Time frames and methods for assessment of outcomes are specified elsewhere.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group: Usual physical activity habits (No Intervention): The participants will receive a wrist-worn activity tracker (Garmin VívoSmart 5) including clear instructions on how to use the tracker and how to connect to a software (Fitrockr). We ask the participants to wear the tracker 24/7 during the period they are trying to conceive and during the first trimester of their pregnancy if they conceive within 12 months to measure physical activity. Participants in the control group will not receive any PA feedback.
  Participants are advised to maintain their usual activity habits.
- Intervention group: Changing physical activity habits (Experimental): The participants will receive a wrist-worn activity tracker (Garmin VívoSmart 5) including clear instructions on how to use it. They will be asked to wear the tracker 24/7 during the period they are trying to conceive plus the first trimester of their pregnancy. They will receive information material on the Danish national guidelines on PA, health benefits from PA, and suggestions on how to reduce sedentary behavior and increase daily activity. Based on the current PA level, they are asked to set personal goals to meet the PA recommendations and to split up sedentary behavior. They will receive a phone call two and five weeks after they received the activity tracker, to stimulate the participant's motivation to be physically active, to set goals for maintaining or increasing PA and to facilitate a revision of the goals if needed.
  The conversations will be inspired by motivational interviewing and the principles of this motivational technique.
  Interventions: Behavioral: Use of activity trackers and motivational conversations to enhance focus on physical activity among women trying to conceive.

INTERVENTIONS:
Behavioral: Use of activity trackers and motivational conversations to enhance focus on physical activity among women trying to conceive. — All participants will receive a wrist-worn activity tracker (Garmin VívoSmart 5) which will be connected with an application, Fitrockr. Data from the devices will be linked to data from the Snartforældre-questionnaires. The participants are asked to wear the tracker 24/7 during preconception and during the first trimester of their pregnancy if they conceive within 12 months.
  Participants will receive information material and be asked to set goals for their PA level. To follow-up on the goal setting, they will receive two phone calls, where the conversations will be inspired by motivational interviewing.
  Arms: Intervention group: Changing physical activity habits

SUMMARY:
Physical activity in both the preconception period and during pregnancy may enhance the probability of getting pregnant and reduce the risks of complications during pregnancy. Adults, including pregnant women without complications, are recommended to be physically active for at least 30 minutes per day to maintain physical and mental health. Nonetheless, many women reduce their level of exercise during early pregnancy.

With this project, we will test the effectiveness of receiving motivational counseling on physical activity (PA) among women trying to conceive and during the first trimester of the pregnancy if they conceive. We will further investigate whether PA is associated with fecundability, spontaneous abortion (SAB) and other birth outcomes, i.e., gestational diabetes, preeclampsia, and birth weight.

DETAILED DESCRIPTION:
Infertility, defined as the failure to achieve pregnancy after 12 months of regular unprotected sexual intercourse, and spontaneous abortion (SAB) are significant public health problems, affecting up to 20% of reproductive age couples in the Western World. A large proportion of couples seek fertility treatment, which is not only an economic burden for the society, but also associated with adverse health effects among infertile couples. The causes of both infertility and SAB are multifactorial and identification of modifiable risk factors is an important public health goal.

According to the Danish Health Authority, adults are recommended to be physically active for at least 30 minutes per day, to undertake muscle-strengthening activities on two or more days per week and to reduce sedentary time. The same applies for pregnant women without complications. However, only 15-38% of pregnant women adhere to the recommendations for PA and many women reduce their level of exercise during early pregnancy compared with pre-pregnancy. Yet, maternal health in both the preconception period and during pregnancy is critical to avoid complications during pregnancy and for the long-term health of mother and child.

We therefore aim to investigate the association between PA, fecundability (i.e., the average per-cycle probability of conception), and SAB. An efficient web-based infrastructure to recruit, follow, and collect comprehensive data has already been developed. In the ongoing prospective cohort study, SnartForældre.dk (SF), we investigate fecundability and SAB according to demographic, behavioral, environmental, and medical factors and have enrolled more than 10,000 women and 1,700 of their male partners who are trying to conceive without fertility treatment.

In the present SF sub-study, SnartForældre.dk/Aktivitet, we aim to conduct a two-armed randomized controlled trial with 500 women included, to investigate the effectiveness of receiving motivational counseling on physical activity (PA) among women trying to conceive and during the first trimester of the pregnancy if they conceive. We will further investigate whether PA is associated with fecundability, spontaneous abortion (SAB) and other birth outcomes, i.e., gestational diabetes, preeclampsia, and birth weight. As we will be able to combine self-reported data, objectively measured data on PA, and high-quality Danish registry data, we have a unique possibility to evaluate the impact of PA on fecundability and SAB, as well as other pregnancy complications and birth outcomes, in a way that is hardly possible in any other country.

The study will provide important knowledge that will be of interest for the scientific world, health professionals, and for couples who suffer from infertility or experience SABs.

ELIGIBILITY:
Inclusion Criteria:

* Female
* 18-49 years
* In a relationship with a male partner
* Trying to conceive

Exclusion Criteria:

* Using birth control
* Receiving fertility treatment
* Have been trying to conceive for more than six months

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — To participate in the study, the participants must be females and registered with a Danish Civil Registration Number as a female. Participants must be trying to conceive with a male partner without fertility help.
Enrollment: 530 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Physical activity | From randomization to end of study or censoring event, no more than 15 months
  Physical activity will be objectively measured continuously (24/7) using wrist-worn activity trackers with triaxial accelerometry.
Time to pregnancy (TTP) | From baseline until they report a pregnancy or a censoring event (12 cycles of follow-up, cessation of pregnancy attempt, initiation of fertility treatment, withdrawal or loss to follow-up), no more than 12 months
  TTP will be estimated by using variables from baseline and follow-up questionnaires. In each follow-up questionnaire, women report the date of the first day of their last menstrual period (LMP), whether they are currently pregnant, and whether they experienced any other pregnancies (SAB, induced abortion, or ectopic pregnancy) since their last questionnaire. For irregularly cycling women, we estimate cycle length based on baseline LMP date, expected date of next menses, and LMP recorded during follow-up.
Spontaneous abortion | From reported pregnancy until spontaneous abortion or censoring event (≥22 weeks' gestation, emigration, medically induced abortion or ectopic pregnancy), no more than 22 weeks from study entry
  Spontaneous abortion (SAB), defined as an intrauterine pregnancy loss before week 22 of gestation, will be identified from both bimonthly follow-up questionnaires and registries. In follow-up questionnaires, women report if they have had a pregnancy loss since the date of the most recent completed questionnaire as well as the date of loss and the gestational age at loss. Using the civil registration number (CPR), we will retrieve data from the Danish National Patient Registry (DNPR) and the Danish Medical Birth Registry (DMBR) to identify SABs and induced abortions occurring after the baseline enrollment date. For SABs identified from both registry and questionnaire data, we will use data from the DNPR (based on early ultrasound fetometry or LMP) to ascertain the time of SAB.

OTHER OUTCOMES:
A process evaluation assessing the implementation and mechanisms of impact of the SnartForældre.dk/Activity intervention | From inclusion to end of study or censoring event, no longer than 2 years
  A mixed methods process evaluation using the UK Medical Research Council's process evaluation framework to assess implementation (reach, fidelity, and dose) and mechanisms of impact of the intervention. We will collect data through motivational conversations and activity trackers, which provide both qualitative and quantitative insights.
  Through motivational conversations with participants, we will capture their experiences, challenges, and suggestions regarding the intervention. This qualitative feedback helps us understand context-specific issues.
  Data from activity trackers will offer objective measures of participant behavior and engagement with the intervention, allowing us to identify trends, such as compliance and changes in activity levels, that may indicate whether the intervention is being followed as intended.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Sofie Dam Laursen, cand.scient, ph.d.,, Study Chair — Department of Clinical Epidemiology, Aarhus University
Locations (1):
- Department of Clinical Epidemiology, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Study website — https://snartforaeldre.dk/

DOCUMENTS (1):
  • Statistical Analysis Plan (2024-11-11): https://cdn.clinicaltrials.gov/large-docs/12/NCT06705712/SAP_000.pdf